CLINICAL TRIAL: NCT01749592
Title: Hemispheric Dominance in Single-sided Postlingual Deafness and Changes / Plasticity Induced by Cochlear Implants
Brief Title: Single-sided Deafness and Cochlear Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0034
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Sensorineural Hearing Loss (Disorder)
Keywords: hearing loss; cochlear implant; PET; EEG; MEG
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear Implant (Experimental): Surgical Implantation of a Cochlear Implant
  Interventions: Device: cochlear implant

INTERVENTIONS:
Device: cochlear implant — Surgical implantation of a cochlear implant device

SUMMARY:
* As the left and right hemisphere are specialized for different auditory tasks, the proposed study aims at demonstrating different consequences of right or left-sided deafness for the affected individual.
* Furthermore, the question should be answered if auditory deficits and plastic changes can be partially reversed by cochlear implantation of the deaf ear.
* Multicenter, prospective, open, non-randomized clinical trial with 5 patients with right-sided and 5 patients with left-sided sensineural deafness.
* Pre-operative: Audiometry, Sound Localization Audiometry, PET, EEG/MEG
* Comparison of pre-operative investigations with 10 healthy subjects (age and gender matched control group)
* Cochlea implantation
* Follow-up Visits at 3, 6, 9 and 12 month post-operative: Audiometry, Sound Localization Audiometry, PET, EEG, Questionnaires
* Trial with medical device

DETAILED DESCRIPTION:
Postlingual single-sided deafness (SSD) is a type of hearing impairment with normal hearing in one ear and severely impaired hearing in the other ear. The condition induces multiple changes of neural plasticity in central auditory pathways. One manifestation reflects an increased common activation of the contralateral and ipsilateral pathways after stimulation of the normal hearing ear which is correlated with an increased activity between the contralateral and ipsilateral hemispheres. As the left and right hemisphere are specialized for different auditory tasks, the proposed study aims at demonstrating different consequences of right or left-sided deafness for the affected individual. Furthermore, the question should be answered if auditory deficits and plastic changes can be partially reversed by cochlear implantation of the deaf ear. It is assumed that some changes induced by SSD can be detected only by reversal through a cochlear implant.

ELIGIBILITY:
Inclusion criteria: • Patients with acquired single sided sensorineural deafness due to cochlear damage.

* Age: 18-70 years old.
* Onset of SSD within 6 months to 10 years before Study inclusion.
* Normal hearing on the contralateral ear (Hearing thresholds 0.125-2 kHz 25 dB HL or better, 4-8 kHz 35 dB HL or better, 100% speech discrimination at 80 dB SPL).
* Regular middle ear function on the hearing ear.
* Regular structure of the cochlea and the cochlear nerve (as demonstrated by MRI, MRI scans are included in the basic assessment of SSD and are no study-specific investigations).
* Fluency in the German language.
* Subject is willing to comply with all study requirements.
* Impairment in daily life as a consequence of SSD (communication problems, annoyance by tinnitus perception).
* Subject is not participating in another ongoing research study related to the SSD.
* Subject does not have unrealistic expectations, regarding the outcome of the intervention.
* Subject has had a trial with conventional acoustic measures in SSD (CROSS, BAHA).

Exclusion criteria: • Uncertainty of correct diagnosis of SSD.

* Retrocochlear cause of SSD (Deafness due to lesions of the acoustic nerve or central auditory pathways).
* Active middle ear infections.
* Ossification of the cochlear that prevents electrode insertion.
* Tympanic membrane perforation.
* Psychiatric comorbidities such as depression or cognitive deficits.
* Severe coexisting illness with a medium survival of less than 5 years.
* Exposure to radiation with a cumulative effective dose of 5 mSV within the last 5 years (including the ongoing year).
* Increased risk profile for general anesthesia due to cardiovascular comorbidity.
* Metallic implants constituting an exclusion criterium for MEG procedures of the brain.
* Pregnancy (a pregnancy test will be performed in women in the reproductive age group before study enrolment and before postoperative PET scan) and lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2018-01 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Audiometry | up to12 months after invention
  Pure tone audiometry Speech audiometry Sound localization in both quiet and noise

SECONDARY OUTCOMES:
PET scan | 9 months after intervention
  [15O] H2O Positron emission tomography (PET) is performed. The comparison of baseline PET scans and stimulated PET scans will demonstrate task related changes in brain activity

OTHER OUTCOMES:
EEG | 3, 6 and 12 months after intervention
  Resting state EEG and EEG with acoustic paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kleinjung, MD, Principal Investigator — University Hospital Zurich, Division of Otorhinolaryngology ORL
Locations (1):
- University Hospital Zurich, Division of Otorhinolaryngology ORL, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peter N, Treyer V, Probst R, Kleinjung T. Auditory Cortical Plasticity in Patients with Single-Sided Deafness Before and After Cochlear Implantation. J Assoc Res Otolaryngol. 2024 Feb;25(1):79-88. doi: 10.1007/s10162-024-00928-3. Epub 2024 Jan 22. PMID 38253897
- [Derived] Peter N, Kleinjung T, Probst R, Hemsley C, Veraguth D, Huber A, Caversaccio M, Kompis M, Mantokoudis G, Senn P, Wimmer W. Cochlear implants in single-sided deafness - clinical results of a Swiss multicentre study. Swiss Med Wkly. 2019 Dec 27;149:w20171. doi: 10.4414/smw.2019.20171. eCollection 2019 Dec 16. PMID 31880806